CLINICAL TRIAL: NCT04775628
Title: Forces and Translation Distance During an Inferior Glide of the Shoulder in Healthy Subjects Measured With the Novel Pliance Glove and Ultrasound Imaging
Brief Title: Forces and Translation Distance During an Inferior Glide of the Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Rob Sillevis, (Other)
Collaborators: Mitchell Todd (Unknown); J.P Speare (Unknown); Eric Shamus (Unknown); Arie van Duijn (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Rob Sillevis,, Assistent Professor, Florida Gulf Coast University
Organization: Florida Gulf Coast University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-015
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2021-02

CONDITIONS: Asymptomatic Condition
Keywords: Manipulation force; Glenohumeral joint; Musculoskeletal Ultrasound Imaging
MeSH Terms: conditions — Asymptomatic Diseases

STUDY DESIGN:
Intervention Model Description: Within subject design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- inferior glide (Experimental): Inferior glide of the right humerus till no motion is visual on the imaging
  Interventions: Procedure: Inferior glide humerus in GH joint

INTERVENTIONS:
Procedure: Inferior glide humerus in GH joint — Supine inferior glide GH joint

SUMMARY:
This study evaluates the force and translation distance in the GH joint during a manual inferior glide of the humerus.

DETAILED DESCRIPTION:
There has been limited research on how the variance of force affects MT outcomes and what the best practices of MT should be. No specific force threshold necessary to achieve a predetermined translational distance within the joint has been quantified within the literature. The purpose of this study was to quantify the amount of force necessary to perform an inferior glide to the glenohumeral joint and reach to end-range. A secondary aim was to determine the impact of co-variables, such as gender, height, weight, and age, on the amount of force required to translate the humeral head within the glenohumeral joint. Musculoskeletal Ultrasound imaging using the GE LogiQe was used to measure the translation of the humeral head. The manipulation force was measured using the Novel Pliance Glove device and software.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Able to read the English language fluently

Exclusion Criteria:

* a history of injury of the right shoulder
* right shoulder surgery
* presence of shoulder pain
* comorbidities affecting natural ROM within the dominant shoulder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Translation | 5 minutes
  Measured in mm using MSK Ultrasound
Force measure | 5 minutes
  Force measure during inferior glide using Novel Pliance Glove

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Gulf Coast University, Fort Myers, Florida, United States

IPD SHARING:
Plan to Share IPD: No